CLINICAL TRIAL: NCT00633802
Title: Low-Dose Risperidone Treatment for Subjects Suffering From Borderline Personality Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Miki Bloch, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-089
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Borderlone Personality Disorder
Keywords: Risperidone; Borderlone Personality Disorder
MeSH Terms: interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: Risperidone
- 1 (Experimental)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — 1 mg/d risperidone for 10 weeks or placebo

SUMMARY:
Personality disorders are life-long maladaptive behavioral patterns. Borderline personality disorder (BPD) is the leading personality disorder encountered in clinical settings, often associated with tremendous distress. It is characterized by impulsivity, emotional lability, unstable interpersonal relationships, with particular sensitivity to abandonment. BPD patients are prone to self destructive behaviors and all too frequently attempt suicide. When in emotional turmoil, persons with BPD may also develop brief, transient psychotic states.

Psychotherapy for BPD is a common treatment option, but it requires considerable time and specific personnel training, and is therefore not always feasible. Medical treatment is an efficacious alternative, however there is no concensus on drug selection. Some experts have suggested that medical treatment should be selected individually according to the subject's dominant clinical symptom. Several psychopharmacological groups have been proposed: Antidepressants, mood stabilizers, and several novel antipsychotic drugs. The latter are particularly promising since they may produce symptomaic improvement with fewer adverse effects. Risperidone has been shown in a few preliminary studies to be promising in the treatment of various BPD symptoms, but no controlled study has tested it yet. We propose to test the efficacy of risperidone in the treatment of BPD in a double-blind crossover design using both clinical and phsysiological measure.The main hypothesis is that risperidone will be efficient in alleviating BPD core and secondary symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Women with Borderline PD according to DSM-IV
2. Signed informed consent.
3. Age 18-45.

Exclusion Criteria:

1. Psychotic disorders (past or present).
2. Substance or alcohol related disorders (past or present).
3. Current major depressive episode.
4. Suicidal risk.
5. History of head trauma, which caused loss of consciousness or peritraumatic amnesia or necessitated hospitalization.
6. Any known psychiatric or general medical condition currently requiring specific medical attention.
7. Current treatment with any antipsychotic, antidepressant drugs or mood stabilizers.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-04; Primary Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Improvement Scale | 0, 1, 5, 10 week

CONTACTS AND LOCATIONS:
Overall Officials: Miki Bloch, Ph.D., Principal Investigator — The Tel-Aviv Sourasky Medical Center
Locations (1):
- Psychiatric Service, Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174